CLINICAL TRIAL: NCT01037543
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Escalating Single-Dose Study to Evaluate the Safety, Tolerability, and PK of HM10460A (HNK460) When Administered Subcutaneously to Healthy Adult Japanese and Caucasian Subjects.
Brief Title: Safety and PK of HM10460A (HNK460) in Healthy Adult Japanese and Caucasian Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-HM10460A-101
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
MeSH Terms: interventions — eflapegrastim; pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 1.1 mcg/kg of HM10460A, placebo, or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta
- Cohort 2 (Experimental): 3.3 mcg/kg HM10460A, placebo or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta
- Cohort 3 (Experimental): 10 mcg/kg of HM10460A, placebo, or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta
- Cohort 4 (Experimental): 30 mcg/kg of HM10460A, placebo, or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta
- Cohort 5 (Experimental): 90 mcg/kg or HM10460A, placebo, or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta
- Cohort 6 (Experimental): 270 mcg/kg of HM10460A, placebo, or Neulasta
  Interventions: Drug: HM10460A or placebo or Neulasta

INTERVENTIONS:
Drug: HM10460A or placebo or Neulasta — Single SC injection of the appropriate dose of drug ranging from 1.1 mcg/kg to 270 mcg/kg.
  Other Names: LAPS-G-CSF

SUMMARY:
Study Design

* Randomized, double-blind, placebo-controlled, escalating single-dose design.
* Six ascending dose cohorts
* In each cohorts, subjects will be randomized to receive a single dose of HM10460A, placebo (negative control), or Neulasta® (positive control).
* Primary Objective
* to assess the safety and tolerability of single escalating subcutaneous doses of HM10460A in healthy adult Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
Secondary objectives:

* to assess the pharmacokinetics (PK) of a single subcutaneous dose of HM10460A.
* to compare the PK of HM10460A in Japanese and Caucasian subjects.
* to assess the relationship between the serum concentration of HM10460A and absolute neutrophil count (ANC).
* to assess the relationship between the serum concentration of HM10460A and CD34+ cell counts in the blood.
* To assess the immunogenicity potential of HM10460A by measuring binding antibodies (bAb) and neutralizing antibodies (nAb) to HM10460A and native G-CSF following a single subcutaneous dose of HM10460A.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 18 - 29.9 kg/m2
* have not used tobacco or nicotine containing products for at least 3 months prior to dosing
* be able to remain abstinent throughout the study.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
* positive urine drug/alcohol testing
* Positive for HIV, HBsAg, HCV ab
* History of anaphylactic reaction to medicine or environmental exposure

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety data, including physical examinations (to include injection site reactions and splenic evaluations), laboratory evaluations, ECGs, vital signs assessments, and adverse effects (AEs). | Time points where appropriate.
Samples for immunogenicity | Days -1, 15, 22, and 42.

SECONDARY OUTCOMES:
PK parameters measured from Serum and Urine samples. | Serum samples: pre-dose, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 hrs, Days 4, 5, 6, 7, 11, 15, and 22. / Urine Samples: 0 - 6, 6 - 12, 12 - 24, 24 - 36, and 36 - 48 hours post-dose.
Calculation of ANC and CD34+ cell counts. | pre-dose, 24 and 48 hours post-dose, Days 4, 5, 6, 7, 11, 15, and 22.

CONTACTS AND LOCATIONS:
Overall Officials: Hanmi Clinical, Principal Investigator — California
Locations (1):
- California City, California, United States

REFERENCES:
- [Derived] Jeon Y, Lee N, Baek S, Choi J, Jhee S, Lee H. A Randomized, Double-Blind, Placebo- and Active-Controlled, Escalating Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Profiles of Subcutaneous Eflapegrastim in Healthy Japanese and Caucasian Subjects. Drugs R D. 2022 Mar;22(1):71-87. doi: 10.1007/s40268-021-00379-8. Epub 2022 Jan 6. PMID 34993933